CLINICAL TRIAL: NCT03513315
Title: Heat Emergency Awareness and Treatment (HEAT): A Cluster Randomized Trial to Assess the Impact of a Comprehensive Intervention to Mitigate Humanitarian Crisis Due to Extreme Heat in Karachi, Pakistan
Brief Title: Heat Emergency Awareness and Treatment (HEAT)
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Aga Khan University (Other); Aman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00089663
Record Dates: First submitted 2018-04-12; First posted 2018-05-01 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Heat Illness; Heat Stroke; Heat Exhaustion; Heat Exposure; Heat Syncope, Sequela; Heat Collapse; Heat; Heat Stroke and Sunstroke
Keywords: Heat-related illnesses; Heat Illnesses; Community based interventions; heatwave; Pakistan; emergency preparedness; emergency medicine; heat stroke; heat exhaustion; urban health
MeSH Terms: conditions — Heat Stress Disorders; Heat Stroke; Heat Exhaustion; Sunstroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Community Clusters (Experimental): For the community-based arm of the study, 16 clusters will be randomized into intervention and control groups. Those in the intervention group will receive implementation of community-based Home Heat Bundle. This Bundle includes education from community health workers on the signs and symptoms of heat-related illness, how to prevent the illness, and when to seek treatment. In addition, the intervention group will receive SMS messaging with information about heatwaves. The education and Short Message Service (SMS) messaging will occur in March and April via meetings in households and in public spaces. There will be a total of 40 activities, each lasting approximately two hours.
  Interventions: Behavioral: Implementation of Community-based Home Heat Bundle
- Control Community Clusters (Experimental): Eight community clusters of 1000 population each where regular community-based healthcare services will be provided without focused interventions on identification and management of heat-related illnesses. These clusters will receive regular community healthcare provision.
  Interventions: Behavioral: Regular Community Healthcare provision

INTERVENTIONS:
Behavioral: Implementation of Community-based Home Heat Bundle — This community-based intervention include a set of educational materials to increase awareness about heat-related illness and prevention with the intention of reducing the incidence of heat-related and reducing mortality associated with heat-related illness. Materials used in this intervention will include posters, brochures, in-person training, and SMS messaging.
  Arms: Intervention Community Clusters
Behavioral: Regular Community Healthcare provision — The community will get regular community health workers visit without the focus community mobilization and education on heat-related illnesses.
  Arms: Control Community Clusters

SUMMARY:
Investigators propose an intervention trial of a comprehensive education and treatment bundle designed to reduce morbidity and mortality associated with heat-related illness for low resource settings. Two set of interventions will be developed each for emergency department and for community/home. These interventions will be developed by an internal expert group and will be customized and implemented at the home and emergency department (ED) levels, will include evidence-based educational training guidelines for ED health providers as well as educational messages targeting home and community in Karachi, Pakistan.

DETAILED DESCRIPTION:
This study consists of a community-based and hospital-based components. The community-based study is a prospective two-arm cluster randomized controlled trial and will be implemented in 16 clusters of 1000 people located in the most central neighborhood (called "mohalla") of a Union Council. Minimum required sample size is 7120 in each group, which requires 890 subjects in each of the 16 clusters. Calculations are based on achieving 80% power to detect a difference between the group proportions of 20% from the baseline.

For the hospital component, four major hospitals will be randomized to receive operations and clinical capacity building on management of heat emergencies. The hospital sample size is limited by the availability of hospitals and their uneven distribution which are not linked to union councils in the district.

The primary outcome in the investigators' study is the frequency of emergency admissions to the hospital with all-cause mortality as a secondary outcome.

A community-based and hospital-based protocols and training materials will be developed and will serve as the intervention in this study. These will focus on education about recognizing the signs of symptoms of heat-related illness and proper response and treatment based on local resources.

Data collection will be done at baselines and post-intervention. In the community data on demographics and household characteristics will be collected. Additionally, data on deaths in households will be collected. Changes in knowledge, attitudes, and practices will be measured using a Knowledge, Attitudes, and Practices (KAP) survey pre- and post-intervention.

In the hospital, data collection will focus on emergency department admissions, visits, mortality, and heat index. Changes in physician knowledge will be measures with a KAP survey pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency departments in Karachi who present with suspected heat stroke/heat exhaustion and basic information about their presentation and treatment will be obtained in the ED for May-July.
* Community households in "Korangi District"
* Physicians/Nurses working in the emergency department of study hospital sites

Exclusion Criteria:

* When a family refused to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16973 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Emergency Department visits | 3 months
  Total number of individuals requiring visit to an emergency department during the study period

SECONDARY OUTCOMES:
Total number of deaths (due to any cause) | 3 months
  Total number of deaths in the community during the study period
Hospital admissions | 3 months
  Total number of hospital admissions due to any cause during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Junaid A Razzak, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Pakistan (2):
  - Aga Khan University, Karachi
  - The Aman Foundation, Karachi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Razzak JA, Agrawal P, Chand Z, Quraishy S, Ghaffar A, Hyder AA. Impact of community education on heat-related health outcomes and heat literacy among low-income communities in Karachi, Pakistan: a randomised controlled trial. BMJ Glob Health. 2022 Jan;7(1):e006845. doi: 10.1136/bmjgh-2021-006845. PMID 35101860